CLINICAL TRIAL: NCT05985980
Title: The Effects of Menstrual Cycle Phase on Exercise Treadmill Test Results in Premenopausal Women
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mehmet Agirbasli MD, Medical Doctor, Professor of Cardiology, Istanbul Medeniyet University
Other Study IDs: 2023/0129
Record Dates: First submitted 2023-07-18; First posted 2023-08-14 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Menstrual Cycle; Exercise Treadmill

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ETTs will be performed at the early and late follicular phases in premenopausal women: The study population consists of premenopausal women who applied to the outpatient clinic with chest pain between February 2023 and July 2023. ETTs are planned as part of the routine clinical workup. The history of the patient's menstrual cycle is obtained in detail. The early and late follicular phases are determined from the history. Two separate ETTs are performed on each patient. The early follicular phase ETT is planned on the 3rd day of menstrual bleeding, while the menstrual bleeding continues. The late follicular phase ETT is planned on the 3rd day after the menstrual bleeding ends. Hormone levels are measured before each ETT to ascertain the phase of the menstrual cycle.
  Interventions: Diagnostic Test: Exercise Treadmill Test (ETT)

INTERVENTIONS:
Diagnostic Test: Exercise Treadmill Test (ETT) — The study population consists of premenopausal women who applied to the outpatient clinic with chest pain. ETT is ordered as a routine diagnostic workup. Two ETTs are performed on each participant. The early follicular phase ETT is planned on the 3rd day of menstrual bleeding, while the menstrual bleeding continues. The late follicular phase ETT is planned on the 3rd day after the menstrual bleeding ends. Hormone levels are measured before each ETT to ascertain the phase of the menstrual cycle.

SUMMARY:
False positive results are commonly observed in women after exercise treadmill test (ETT). The effects of menstrual cycle on the results of ETT in premenopausal women have not been clearly defined. Primary purpose of the study is to investigate the biological causes of false positive test results in the ETT in premenopausal women. Estrogen is known to have direct vasodilatory effects on coronary arteries. The early and late follicular phases of the menstrual cycle are characterized by low and high estrogen levels, respectively. The early follicular phase starts on the first day of the menstrual cycle and ends when estrogen begins to increase. It is characterised by increasing luteinizing hormone (LH) and follicle stimulating hormone (FSH) and low estrogen levels. The estrogen levels increase several folds in the late follicular phase. The hypothesis of the study is that ETT results will change at the early and late follicular phases of the menstrual cycle in premenstrual women. Premenopausal women between the ages of 20-55 years, who apply to the cardiology outpatient clinics of Göztepe City Hospital with chest pain. Patients who are ordered to have an ETT will be included in the study. ETT will be performed separately during the early and late follicular phases of the menstrual cycle.

DETAILED DESCRIPTION:
General Hypothesis:

False positive results are commonly observed in women after exercise treadmill test (ETT). The studies report severe variability in the sensitivity and specificity of ETT in detecting significant coronary artery disease (CAD). Sensitivity ranges from 23% to 100% and specificity ranges from 17% to 100%. ETT utilizes electrocardiography (ECG) along with heart rate (HR) and blood pressure (BP) monitoring during exercise, typically involving a treadmill. The major finding of ETT is the ST segment deviation from the baseline. False positive stress ECGs are common especially in premenopausal women, limiting the specificity of the test.

Menstrual periods can cause biological variability in ETT in premenopausal women. The menstrual period is divided into phases: early follicular (days 1-5), late follicular (days 6-12), ovulation (days 13-15), early luteal (days 16-19), mid-luteal (days 20-23) and late luteal phases (24-28 days). Early follicular phase is characterized by low estrogen and low progesterone, late follicular phase is characterized by low progesterone and high estrogen. Mid-luteal phase is characterized by high progesterone and high estrogen levels. Early and late follicular phases of the menstrual cycle in women demonstrate nearly 4 fold differences in estrogen levels. The menstrual period phase affects thermoregulation and physical working capacity in women. Estrogen has protective and vasodilatory effects on the cardiovascular system. With the discovery of high sensitive cardiac troponins (hs-cTn), minute changes of hs-cTn have become detectable.

The effects of menstrual periodic changes on the results of exercise treadmill test in premenopausal women have not been clearly defined. Primary purpose of the study is to investigate the biological causes of false positive test results in the treadmill exercise test in premenopausal women. Estrogen is known to have direct vasodilatory effects on coronary arteries. Early and late follicular phases of the menstrual cycle are characterized by low and high estrogen levels, respectively. The Early Follicular Phase starts on the first day of the menstrual cycle and ends when oestradiol begins to increase. It is characterised by increasing LH and FSH and constant low levels of oestradiol. The late follicular phase starts with the increase in oestradiol and ends at its preovulatory peak. False positive stress ECGs are commonly reported especially in premenopausal women, limiting the specificity of the ETT. Studies demonstrated that HR adjustment of in exercise-induced ST segment depression using the ST/HR slope or ST/HR index could improve the sensitivity and specificity of ETT.

The hypothesis of the study is that ETT results and hs-cTnT release after ETT will change at the early and late follicular phases in premenstrual women.

2. STUDY ENDPOINTS

The major finding of ETT is the ST segment deviation from the baseline. The ST segments are evaluated 60-80 ms after the J point. ECG positive ETT result was defined as ≥ 1 mm (0.1 mV) horizontal or downsloping ST depression in at least 3 consecutive beats.

Chest pain or inadequate hemodynamic response during ETTs are considered clinically positive ETT result. Tests that do not meet these criteria but show ST segment changes or had low diagnostic value due to baseline ECG changes are considered indeterminate ETT results.

Automated measurements and mathematical calculations are recorded in the ETT system (General Electronic GE Healthcare T2100-ST Treadmill & CASE 6.73 Stress Test System).

ETT results are evaluated by 2 different cardiologists and categorized as positive/indeterminate/negative ETT results.

Hs-cTn is measured before and 15 minutes after ETT.

Indices of ST/HR slope and the ST/HR index were reported automatically by the General Electronic GE Healthcare T2100-ST Treadmill & CASE 6.73 Stress Test System device. The primary endpoint in the study was the ST/HR index. The secondary endpoints were ST/HR slope, maximum ST segment depression (mm), maximum exercise capacity, and the change in estrogen levels between the early and late follicular phases of the menstrual cycle. The study will also compare hs-cTnT before and after ETT.

Primary endpoint:

ST/HR index during ETTs at the early and late follicular phases of the menstrual cycle (µV/beats per minute (bpm))

Secondary endpoints:

1. Change in maximal exercise capacity with exercise and menstrual cycle (METs score)
2. maximum ST segment depression (mm)
3. ST/HR slope (µV/beats per minute (bpm))
4. The change in high-sensitive cardiac troponin T after ETT (ng/L)
5. Hormone levels (estrogen) at the early and late follicular phases of the menstrual cycle

3. STUDY DESIGN The study is performed in the cardiology clinics of a tertiary care training hospital. The study is approved by the local ethics committee (number 2023/0129 on 22/02/2023).

Study Population:

The study population consists of premenopausal women who applied to the outpatient clinic with chest pain between February 2023 and July 2023. Patients report that they have a regular menstrual cycle. Written informed consent is obtained from the patients.

All patients have transthoracic echocardiography. Echocardiography demonstrates normal left ventricular systolic and diastolic function. Echocardiography does not show wall motion abnormality or significant valvular heart disease.

All patients are evaluated for cardiovascular risk. Risk factors such as hypertension, diabetes mellitus, cigarette smoking, hyperlipidemia, family history of CAD, and drug use are questioned. Cardiovascular risk factors are defined as follows. Hypertension is defined as a persistent elevation in office systolic BP ≥140 and/or diastolic BP ≥90 mmHg, or a 24-hour ambulatory BP monitor average of ≥130/80, or requirement of chronic use of antihypertensives. Hyperlipidemia is defined as elevated total cholesterol (>240 mg/dl), low-density lipoprotein cholesterol (LDL-C) (>160 mg /dl), triglycerides > 150 mg/dl, high-density lipoprotein cholesterol (HDL-C) (< 50 mg /dl). Cigarette smoker is defined as having smoked at least 100 cigarettes in life time. Type 2 diabetes mellitus is defined as fasting plasma glucose (FPG) ≥ 126 mg/dL, or 2-hour plasma glucose ≥ 200 mg/dL during a 75-g oral glucose tolerance test (OGTT), or random plasma glucose ≥ 200 mg/dL in a patient with classic symptoms of hyperglycemia, or hemoglobin A1c (HbA1c) ≥ 6.5% (48 mmol/mol). Self-reported family history of premature CAD is defined as having a first-degree relative with premature CAD (men, age <55 years; women, age <65 years).

Menstrual cycle The history of the menstrual cycle of the patient is obtained in detail. The early and late follicular phases are determined from the history.

The early follicular phase ETT is planned on the 3rd day of menstrual bleeding, while the menstrual bleeding continues. The late follicular phase ETT is planned on the 3rd day after the menstrual bleeding ends. Hormone levels are measured before each ETT to ascertain the phase of the menstrual cycle. Two ETTs are performed on each participant.

The duration and regularity of the menstrual cycle, the amount of bleeding, and the number of days the bleeding lasted are noted for each patient. Patients with irregular menstrual cycles, breakthrough bleeding, spotting, gynecological examination, or treatment plan that would disrupt the menstrual cycle are excluded from the study.

The blood sample is taken 30 minutes before the ETT to measure follicular stimulating hormone (FSH), luteinizing hormone (LH), estrogen, progesterone, and hs-cTn. After the test, the patient is allowed to rest for 15 minutes and blood is taken to check the 2nd hs-cTn after ETT.

The inclusion criteria are:

1. Premenopausal female patients with regular menstrual cycles,
2. Ages between 20-55 years,
3. Patients have been seen in the cardiology clinic by a cardiologist for the symptoms of chest pain with a clinical suspicion of angina or angina equivalent.
4. A cardiologist has ordered ETT as a diagnostic test independent of the study protocol
5. Patients can understand and sign the informed consent.

The exclusion criteria are:

1. Women with menopause or menopause-related symptoms or menstrual cycle irregularity or use of hormonal therapy or oral contraceptives, current pregnancy
2. Patients with a history of CAD, secondary or uncontrolled hypertension, valvular heart disease, cardiac arrhythmia or heart failure, pericarditis or myocarditis.
3. Left ventricular hypertrophy on echocardiography, abnormal systolic or diastolic function or wall motion abnormality on echocardiography.
4. History of cancer, stage ≥ 3 kidney failure, liver failure, history of psychiatric illness, history of recent infection.
5. Pre-existing ECG abnormality that would confound the interpretation during the ETT (baseline ECG was considered abnormal ın the presence of the following findings: prolonged QT interval, chamber hypertrophy, alterations in the ST-T waves, any degree of heart block, T-wave abnormalities, premature ventricular contractions (PVCs), right bundle branch block (RBBB), left bundle branch block (LBBB), left or right axis deviation, or any abnormal rhythm other than normal sinus rhythm).
6. Patients who cannot tolerate Bruce protocol in the first ETT.
7. Lack of ability or mental capacity to understand the study.

ELIGIBILITY:
The inclusion criteria are:

1. Premenopausal female patients with regular menstrual cycles,
2. Ages between 20-55 years,
3. Patients have been seen in the cardiology clinic by a cardiologist for the symptoms of chest pain with a clinical suspicion of angina or angina equivalent.
4. A cardiologist has ordered ETT as a diagnostic test independent of the study protocol
5. Patients can understand and sign the informed consent.

The exclusion criteria are:

The exclusion criteria are:

1. Women with menopause or menopause-related symptoms or menstrual cycle irregularity or use of hormonal therapy or oral contraceptives, current pregnancy
2. Patients with a history of CAD, secondary or uncontrolled hypertension, valvular heart disease, cardiac arrhythmia or heart failure, pericarditis or myocarditis.
3. Left ventricular hypertrophy on echocardiography, abnormal systolic or diastolic function or wall motion abnormality on echocardiography.
4. History of cancer, stage ≥ 3 kidney failure, liver failure, history of psychiatric illness, history of recent infection.
5. Pre-existing ECG abnormality that would confound the interpretation during the ETT (baseline ECG was considered abnormal ın the presence of the following findings: prolonged QT interval, chamber hypertrophy, alterations in the ST-T waves, any degree of heart block, T-wave abnormalities, premature ventricular contractions (PVCs), right bundle branch block (RBBB), left bundle branch block (LBBB), left or right axis deviation, or any abnormal rhythm other than normal sinus rhythm).
6. Patients who cannot tolerate Bruce protocol in the first ETT.
7. Lack of ability or mental capacity to understand the study.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients in the pre-menopausal period
Study Population: The study population consists of premenopausal women who applied to the outpatient clinic with chest pain. ETT is ordered as a routine diagnostic workup. Two ETTs are performed on each participant. The early follicular phase ETT is planned on the 3rd day of menstrual bleeding, while the menstrual bleeding continues. The late follicular phase ETT is planned on the 3rd day after the menstrual bleeding ends. Hormone levels are measured before each ETT to ascertain the phase of the menstrual cycle.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sukru Sadık Öner, MD PhD, Study Director — Istanbul Medeniyet University City Hospital Goztepe
Locations (1):
- Istanbul Medeniyet University Hospital, Goztepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results will be published as journal article

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Repeated exercise treadmill tests (ETT) are performed by using the standard Bruce protocol, during early and late follicular phases of menstrual cycle.
Groups:
- All Study Participants Undergo 2 Consecutive Exercise Treadmill Tests (ETT): Exercise treadmill test (ETT) is performed at the early and late follicular phase of the menstrual cycle.
Period: Overall Study
Arm/Group | All Study Participants Undergo 2 Consecutive Exercise Treadmill Tests (ETT)
Started | 47 (47 patients completed the first ETT.)
Completed | 43 (43 patients completed the 1st and 2nd ETT.)
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Exercise Test Results Are Performed at the Early and Late Follicular Phases of Menstrual Cycle.: The study population consists of premenopausal women who applied to the outpatient clinic with chest pain between February 2023 and July 2023. Patients report that they have a regular menstrual cycle. Written informed consent is obtained from the patients. All patients have transthoracic echocardiography. Echocardiography demonstrates normal left ventricular systolic and diastolic function. Echocardiography does not show wall motion abnormality or significant valvular heart disease. All patients are evaluated for cardiovascular risk. The history of the menstrual cycle of the patient is obtained in detail. The early and late follicular phases are determined from the history. The early follicular phase ETT is planned on the 3rd day of menstrual bleeding, while the menstrual bleeding continues. The late follicular phase ETT is planned on the 3rd day after the menstrual bleeding ends. Hormone levels are measured before each ETT to ascertain the phase of the menstrual cycle. Two ETTs are performed on each participant. The duration and regularity of the menstrual cycle, the amount of bleeding, and the number of days the bleeding lasted are noted for each patient. Patients with irregular menstrual cycles, breakthrough bleeding, spotting, gynecological examination, or treatment plan that would disrupt the menstrual cycle are excluded from the study.
  The exercise treadmill tests are performed at early and late follicular phases of menstrual cycle for every participant of the study.
Arm/Group | Exercise Test Results Are Performed at the Early and Late Follicular Phases of Menstrual Cycle.
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 43
Premenopausal women with chest pain who are ordered to have ETT as part of routine care. [Count of Participants; unit: Participants] | 43

OUTCOME MEASURES:

1. Primary Outcome: ST/HR Index (μV/Bpm)
Description: The ST/HR index (μV/bpm) is automatically generated by the General Electronic GE Healthcare T2100-ST Treadmill & CASE 6.73 Stress Test System at the end of the exercise treadmill test (ETT).
Time Frame: approximately 15 minutes each during the exercise treadmill tests performed at the early and late follicular phases of the menstrual cycle
Population: ST/HR index (μV/bpm) are compared between the ETTs performed at the early and late follicular phases of menstrual cycle.
Measure: Mean (Standard Deviation); unit: μV/Bpm
Groups:
- Early Follicular Phase: Exercise treadmill tests (ETT) are performed at the early follicular phase of menstrual cycle.
- Late Follicular Phase ETT: Exercise treadmill tests (ETT) are performed at the late follicular phase of menstrual cycle.
Arm/Group | Early Follicular Phase | Late Follicular Phase ETT
Number analyzed (Participants) | 43 | 43
μV/Bpm | 1.2 (0.82) | 1.3 (0.59)
Statistical Analysis 1: Comparison: Early Follicular Phase vs Late Follicular Phase ETT; Test type: Equivalence — The null hypothesis is true that the ST/HR index (μV/bpm) ıs similar between the early and late follicular phases; p = 0.521, t-test, 2 sided

2. Secondary Outcome: High-sensitive Cardiac Troponin T (ng/L) After ETT
Description: High-sensitive cardiac troponin T levels (hs-cTnT) are measured by Roche kit before and after the exercise treadmill test both at the early and late follicular phases of the menstrual cycle.
Time Frame: approximately 1 hour each during the exercise treadmill tests performed at the early and late follicular phase of the menstrual cycle
Population: High-sensitive cardiac troponin T (hs-cTnT) levels are compared before and after ETT at the early and late follicular phases of the menstrual cycle.
Measure: Mean (Standard Deviation); unit: nanogram/liter
Groups:
- Hs-cTnT Before and After ETT at the Early Follicular Phase: High sensitive cardiac troponin T (hs-cTnT) levels are measured before and after the exercise treadmill test (ETT) at the early phase of the menstrual cycle.
- Hs-cTnT Before and After ETT at the Late Follicular Phase: High sensitive cardiac troponin T (hs-cTnT) levels are measured before and after exercise treadmill test (ETT) at the late follicular phase of the menstrual cycle.
Arm/Group | Hs-cTnT Before and After ETT at the Early Follicular Phase | Hs-cTnT Before and After ETT at the Late Follicular Phase
Number analyzed (Participants) | 43 | 43
nanogram/liter
  Hs-cTnT before ETT | 3.3 (1.1) | 3.6 (1.4)
  Hs-cTnT after ETT | 3.6 (1.4) | 3.6 (2.5)
Statistical Analysis 1: Comparison: Hs-cTnT Before and After ETT at the Early Follicular Phase vs Hs-cTnT Before and After ETT at the Late Follicular Phase; High-sensitive cardiac troponin T (hs-cTnT) levels before and after ETT at the early and late follicular phases are compared; Test type: Equivalence — High-sensitive cardiac troponin T (hs-cTnT) levels before and after ETT at the early and late follicular phases are compared; p = 0.109, ANOVA

3. Secondary Outcome: Maximal Exercise Capacity (METs Score)
Description: The maximal exercise capacity (METs score) is automatically generated by the General Electronic GE Healthcare T2100-ST Treadmill & CASE 6.73 Stress Test System at the end of the exercise treadmill test (ETT).
Time Frame: as for outcome 1
Population: ETTs are performed at the early and late follicular phases of the menstrual cycle in premenopausal women.
Measure: Mean (Standard Deviation); unit: METS
Groups:
- Early Follicular Phase: Exercise Treadmill Test (ETT) performed at the early follicular phases of menstrual cycle.
- Late Follicular Phase ETT: Exercise Treadmill Test (ETT) performed at the late follicular phases of menstrual cycle.
Arm/Group | Early Follicular Phase | Late Follicular Phase ETT
Number analyzed (Participants) | 43 | 43
METS | 10.0 (1.9) | 10.5 (1.2)
Statistical Analysis 1: Comparison: Early Follicular Phase vs Late Follicular Phase ETT; ETT maximal exercise capacity (METs score) is compared between the early and late follicular phases of menstrual cycle; Test type: Equivalence — ETT maximal exercise capacity (METs score) is compared between the early and late follicular phases of menstrual cycle; p = 0.111, t-test, 2 sided

4. Secondary Outcome: ST/HR Slope (μV/Bpm)
Description: ST/HR slope (μV/bpm) is automatically generated by the General Electronic GE Healthcare T2100-ST Treadmill & CASE 6.73 Stress Test System at the end of the exercise treadmill test (ETT).
Time Frame: as for outcome 1
Population: ETTs are performed at the early and late follicular phases of the menstrual cycle in premenopausal women.
Measure: Mean (Standard Deviation); unit: μV/Bpm
Arm/Group | Early Follicular Phase | Late Follicular Phase ETT
Number analyzed (Participants) | 43 | 43
μV/Bpm | 1.8 (1.2) | 1.7 (0.5)
Statistical Analysis 1: Comparison: Early Follicular Phase vs Late Follicular Phase ETT; ETT ST/HR slope (μV/bpm) is compared between the early and late follicular phases of menstrual cycle; Test type: Equivalence — ETT ST/HR slope (μV/bpm) is compared between the early and late follicular phases of menstrual cycle; p = 0.414, t-test, 2 sided

5. Secondary Outcome: Maximal Horizontal or Down Slope ST Segment Depression (mm) During Exercise Treadmill Test
Description: Maximal horizontal or down slope ST segment depression (mm) is automatically generated by the General Electronic GE Healthcare T2100-ST Treadmill & CASE 6.73 Stress Test System at the end of the exercise treadmill test (ETT).
Time Frame: as for outcome 1
Population: Exercise treadmill tests are performed separately during the menstrual cycle's early and late follicular phases.
Measure: Mean (Standard Deviation); unit: milimeter
Arm/Group | Early Follicular Phase | Late Follicular Phase ETT
Number analyzed (Participants) | 43 | 43
milimeter | 0.13 (0.08) | 0.15 (0.08)
Statistical Analysis 1: Comparison: Early Follicular Phase vs Late Follicular Phase ETT; Maximal horizontal or down slope ST segment depression (mm) during exercise treadmill test is compared between the early and late follicular phases of menstrual cycle; Test type: Equivalence — Maximal horizontal or down slope ST segment depression (mm) during exercise treadmill test is compared between the early and late follicular phases of menstrual cycle; p = 0.062, t-test, 2 sided

6. Secondary Outcome: Estrogen Levels Before the Exercise Treadmill Test.
Description: Estrogen levels are measured 1 hour before the exercise treadmill test (ETT) at the early and late follicular phases of the menstrual cycle.
Time Frame: approximately 1 hour before the exercise treadmill tests performed at the early and late follicular phases of the menstrual cycle
Population: Estrogen levels before the ETT at the early and late follicular phases.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Estrogen Before the ETT at the Early Follicular Phase: Estrogen is measured approximately 1 hour before the exercise treadmill test at the early follicular phases of menstrual cycle.
- Estrogen Before the ETT at the Late Follicular Phase: Estrogen is measured approximately 1 hour before the exercise treadmill test at the late follicular phase of menstrual cycle.
Arm/Group | Estrogen Before the ETT at the Early Follicular Phase | Estrogen Before the ETT at the Late Follicular Phase
Number analyzed (Participants) | 43 | 43
pg/mL | 33.3 [22.3 to 63.3] | 105.0 [64.7 to 209.0]
Statistical Analysis 1: Comparison: Estrogen Before the ETT at the Early Follicular Phase vs Estrogen Before the ETT at the Late Follicular Phase; Test type: Equivalence — Estrogen levels increase at the late follicular phase; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 1 hour during each session.
Groups:
- Exercise Test Results Will be Grouped Based on the Menstrual Cycle.: Exercise treadmill tests will be repeated at a different menstrual cycle phase in premenopausal women (early versus late follicular phase).
Arm/Group | Exercise Test Results Will be Grouped Based on the Menstrual Cycle.
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT05985980/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT05985980/SAP_001.pdf